CLINICAL TRIAL: NCT00637988
Title: A Multicenter, Open-label, Four-way Crossover Study of the Effects of Esomeprazole, Aspirin and Rofecoxib on Prostaglandin (PGE2) Production, Cyclooxygenase-2 Enzyme Activity and PCNA Expression in Patients With Barrett's Esophagus
Brief Title: Barrett's Esophagus - 315 - 3 Way Cross Over
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, Astra Zeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 316; D9612L00057 (Other: AZ)
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Nexium
MeSH Terms: conditions — Barrett Esophagus | interventions — Esomeprazole; Aspirin; rofecoxib

ARMS (4):
- 1 (Experimental): Nexium 40mg
  Interventions: Drug: Esomeprazole
- 2 (Experimental): Nexium 40mg + aspirin
  Interventions: Drug: Esomeprazole; Drug: Aspirin
- 3 (Experimental): Nexium 40mg + Rofecoxib 25 mg
  Interventions: Drug: Esomeprazole
- 4 (Active Comparator): Rofecoxib 25mg
  Interventions: Drug: Rofecoxib

INTERVENTIONS:
Drug: Esomeprazole — 40mg twice daily
  Other Names: Nexium
  Arms: 1; 2; 3
Drug: Aspirin
  Arms: 2
Drug: Rofecoxib — 25mg once daily
  Arms: 4

SUMMARY:
This study evaluates PGE2 production, COX-2 enzyme activity and PCNA expression in Barrett's metaplastic tissue. All patients will have a baseline endoscopy with multiple biopsies. The patients will then be receive four dosing regimens (esomeprazole, esomeprazole and aspirin, esomeprazole and rofecoxib, or rofecoxib alone) consecutively each for a 10 day dosing period, whilst undergoing further follow up endoscopies and multiple biopsies.

ELIGIBILITY:
Inclusion Criteria:

* A biopsy-proven diagnosis of Barrett's esophagus segment length greater than 2cm with no dysplasia or adenocarcinoma.
* Clinically normal laboratory results and physical findings at screening.

Exclusion Criteria:

* A history of esophageal, gastric or duodenal surgery, including antireflux surgery or endoscopic antireflux procedures, except for simple closure of an ulcer.
* Evidence of the following diseases or conditions:
* Barrett's esophagus less than or greater than 2cm that is positive for high grade dysplasia or adenocarcinoma
* Signs and symptoms of gastric outlet obstruction
* Active peptic ulcer disease
* severe liver disease
* Pancreatitis
* Malabsorption
* Active inflammatory bowel disease
* Severe pulmonary, cardiovascular or renal disease
* Impaired renal function or abnormal urine sediment on repeated examinations
* esophageal stricture or active, severe esophagitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2002-04; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Measure PGE production in Barrett's metastatic tissue & determine the reduction from baseline of PGE production would be equivalent on Day 10 in esomeprazole 40mg bid + aspirin treatment compared to esomeprazole 40 mg bid + rofecoxib 25 mg qd treatment | Baseline esophageal biopsies will be taken and thereafter at Day 10 in each treatment period.

SECONDARY OUTCOMES:
To determine in which of the four treatment groups the reduction in the baseline in PGE2 production, COX-2 enzyme activity and PCNA expression in Barrett's metaplastic tissue is the greatest. | Baseline esophageal biopsies will be taken and thereafter at Day 10 in each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca